CLINICAL TRIAL: NCT05919706
Title: The Effect of Motivational Interview Empowered by Mobile Technology on Self Management, Quality of Life and Satisfaction Level in Type 2 Diabetic Patients
Brief Title: Mobile Technology and Motivational Interviewing in Type 2 Diabetes Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inonu University (Other)
Responsible Party: Principal Investigator, Nermin Kılıç Barmanpek, Principal Investigator, Inonu University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: Diabetes Mellitus and Mobile
Record Dates: First submitted 2023-06-13; First posted 2023-06-26 (Actual); Last update posted 2023-06-27 (Actual); Status verified 2023-06

CONDITIONS: Type 2 Diabetes Mellitus; Gaming; Motivational Interviewing; Self-Management; Quality of Life; Mobile Technology
Keywords: Type 2 Diabetes; Self-Management; Quality of Life; Satisfaction; Nursing; Mobile Technology; Gaming; Motivational Interviewing
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Personal Satisfaction | interventions — Patient Education as Topic; Motivational Interviewing

STUDY DESIGN:
Intervention Model Description: This study was conducted as a randomized controlled experimental study with pretest-posttest-follow-up test.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental Group (Experimental): Pre-test data were collected from patients with Patient Information and Follow-up Form, Diabetes Self-Management Scale (DSMQ) and Short Form-36 Quality of Life Scale (SF-36). After the pre-test, a educational program and a game-based mobile technology application were carried out for 4 weeks, 2 days a week at intervals. After the educational program were completed, motivational interviews were conducted once a week for 4 weeks. In this process, it was ensured that the game-based mobile technology application continued. Post-test data were collected with DSMQ and SF-36 at 2 months (8 weeks after the pre-test). After the post-test, the patients were followed up for 4 weeks. After the follow, with the Patient Information and Follow-up Form, DSMQ, SF-36, and the Satisfaction Questionnaire the follow-test data was collected.
  Interventions: Behavioral: Patient Education with Game-Based Mobile Technology and Motivational Interviewing
- Control Group (No Intervention): Pre-test data were collected from patients with Patient Information and Follow-up Form, Diabetes Self-Management Scale DSMQ) and Short Form-36 Quality of Life Scale (SF-36). After the pre-test data were collected, no intervention was applied to the patients for 3 months (12 weeks), except for routine nursing care. Posttest data were collected with DSMQ and SF-36 2 months (8 weeks) after the pretest data. After the last test, the patients were followed up for 4 weeks, and 3 months (12 weeks) after the start of the study, the Patient Information and Follow-up Form (only the parts containing the features related to the disease and metabolic control variables), DSMQ and SF-36 Scale and follow-up test data were collected.

INTERVENTIONS:
Behavioral: Patient Education with Game-Based Mobile Technology and Motivational Interviewing — Education program, game-based mobile technology and motivational interview were applied to the patients in the experimental group. The patients' self-management, quality of life, and satisfaction level scores for the intervention were determined.
  Arms: Experimental Group

SUMMARY:
Type 2 diabetes patients were divided into experimental and control groups. Patients in the control group received regular nursing care, while those in the experimental group received MI, which is empowered by game-based mobile technology. Pre-test, post-test and follow-up test self-management, quality of life and satisfaction levels scores were determined.

DETAILED DESCRIPTION:
A randomized controlled and experimental study design was used to conduct this research on 64 patients with Type 2 DM. Purpose of this study was to explore how motivational interviewing powered by game-based mobile technology affected self-management, quality of life, and satisfaction in Type 2 diabetes patients.

ELIGIBILITY:
Inclusion Criteria:

* Being 18 years or older,
* Having a diagnosis of Type 2 Diabetes Mellitus according to the ADA diagnostic criteria,
* Being on oral antidiabetic and/or insulin therapy,
* Having a smart phone and knowing how to use it,
* Internet connection (to install mobile technology application),
* Not having participated in motivational interviewing (MG) training before,
* Not having vision and hearing problems,
* Not having a communication problem,
* To be able to read, write and speak Turkish,
* Volunteering to participate in the study and continue the study process.

Exclusion Criteria:

* Having a diagnosis of Type 1 and/or Gestational Diabetes Mellitus,
* Having serious health problems that prevent participation in motivational interviewing,
* Using steroid therapy,
* Having complications that may develop in the long term due to diabetes and having advanced retinopathy, neuropathy, amputation history or active foot wound,
* Having mental confusion, having any psychiatric problems and/or using a psychiatric drug,
* Being unwilling to participate in the study and/or not wanting to continue the study process.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2022-10-06 (Actual); Primary Completion 2023-02-03 (Actual); Study Completion 2023-02-03 (Actual)

PRIMARY OUTCOMES:
DSMQ | Last 8 weeks
  The scale is of a four-point Likert type. The scale has 4 sub-dimensions as "Glucose Management, Diet Control, Physical Activity, Health-Care Use" and a total score. The lowest score of the scale is 0 points and the highest score is 10 points. The higher the score, the higher the diabetes self-management.
SF-36 | Last 4 weeks
  The scale consists of 36 items and 8 sub-dimensions. 8 sub-dimensions have 2 summary sub-dimensions as "Physical Health and Mental Health". There is no total score in the scale. A score between 0-100 is evaluated with sub-dimensions (0: Poor Health, 100: Good Health). Low scores on the scale indicate poor health, while high scores indicate good health.

CONTACTS AND LOCATIONS:
Locations (1):
- Bingol State Hospital, Bingöl, Centrer, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
Can be reviewed by other researchers after the study has been published.
Supporting Information: Study Protocol, SAP, ICF, CSR
Time Frame: Data will be shared as long as they are published.
Access Criteria: Publication Page
URL: https://tez.yok.gov.tr/UlusalTezMerkezi/tezSorguSonucYeni.jsp